CLINICAL TRIAL: NCT00194168
Title: Serum Bank for Assessment of Markers of Ectopic Pregnancy
Brief Title: Ectopic Pregnancy Biomarkers
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 705016; RRU002
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Ectopic Pregnancy
Keywords: ectopic pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (Plasma, Serum)
Oversight: Data Monitoring Committee: No

SUMMARY:
In an attempt to simplify the diagnosis of ectopic pregnancy, the researchers will investigate the presence of specific molecular markers of ectopic pregnancy. The quantification of these (and other proteins) will be performed using the Ciphergen Protein Chip system where serum is sampled with a high-throughput system. The patterns of these peaks will be compared for those with a diagnosis of ectopic pregnancy and normal pregnancy. Later goals of the research will be to identify the actual proteins that correspond to the peaks which discriminate between the two clinical entitles. The goal is to identify a unique protein pattern or protein peak to distinguish a normal intrauterine pregnancy from that of an ectopic implanted gestation.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive-aged women
* Currently pregnant based on serum human chorionic gonadotropin level
* Present for care for pregnancy due to vaginal bleeding and/or pelvic cramping
* Final diagnosis of one of the following:

  1. Live intrauterine pregnancy through 14 weeks, diagnosed by ultrasound demonstrating fetal heart motion
  2. Diagnosed ectopic pregnancy
  3. Ultrasound confirmation of a nonviable gestation (less 14 weeks) such as an anembryonic gestation or a fetal demise

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women undergoing treatment for infertility at the University of Pennsylvania Penn Fertility Practice
Sampling Method: Non-Probability Sample
Enrollment: 1306 (Actual)
Dates: Start 2000-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Southern California Women's and Children's Hospital, Los Angeles, California
  - University of Miami, Miami, Florida
  - University of Pennsylvania Reproductive Research Unit, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Barnhart KT, Guo W, Cary MS, Morse CB, Chung K, Takacs P, Senapati S, Sammel MD. Differences in Serum Human Chorionic Gonadotropin Rise in Early Pregnancy by Race and Value at Presentation. Obstet Gynecol. 2016 Sep;128(3):504-511. doi: 10.1097/AOG.0000000000001568. PMID 27500326
- [Derived] Rausch ME, Sammel MD, Takacs P, Chung K, Shaunik A, Barnhart KT. Development of a multiple marker test for ectopic pregnancy. Obstet Gynecol. 2011 Mar;117(3):573-582. doi: 10.1097/AOG.0b013e31820b3c61. PMID 21343760